CLINICAL TRIAL: NCT05202769
Title: Non-Invasive Vital Signs Monitoring (NIVS) Project
Acronym: NIVS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sciberras, Stephen M.D. (Individual)
Collaborators: University of Malta (Other)
Responsible Party: Principal Investigator, Stephen Sciberras, Primary Investigator, Sciberras, Stephen M.D.
Other Study IDs: NIVS
Record Dates: First submitted 2021-12-10; First posted 2022-01-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Hemodynamic Monitoring; Monitoring, Physiologic
Keywords: Non-invasive monitoring; RGB camera; thermal camera

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: 20 healthy volunteers above the age of 18 in a laboratory setting with video clips taken under varying conditions of lighting, distance between the cameras and the participants' faces and with various positions and limb movements involved.
  Interventions: Other: Video filming
- ICU patients: Group/Cohort Description: 20 patients above the age of 18 years and able to provide consent, admitted to the ICU with various underlying conditions and comorbidities. Video clips are taken under varying conditions of lighting, positions and with ongoing care and procedures.
  Interventions: Other: Video filming

INTERVENTIONS:
Other: Video filming — Video clips taken using RGB and thermal imaging cameras under varying conditions of lighting, movement and procedures taking place.
  Other Names: RGB and thermal camera imaging

SUMMARY:
This study is aimed at non-invasive extraction of cardiovascular and respiratory parameters from red-green-blue (RGB) and thermal imaging cameras from patients in the intensive care unit (ICU) setting. The main focus of this study is in assessing the feasibility of implementing such a camera-based system for prolonged monitoring of patients, identifying limiting factors which may interfere with accuracy or practical aspects of the system, and postulating solutions to overcoming these.

DETAILED DESCRIPTION:
Non-invasive monitoring of vital signs is an area that is gaining increasing popularity in clinical practise due to its advantages of increased comfort to patients and reduced risk of transmission of multidrug resistant organisms. This study aims to assess the feasibility of using RGB cameras and thermal imaging cameras for monitoring of heart rate and rhythm and respiratory rate and rhythm in the intensive care setting.

Videos of patients are taken in the ICU of a Maltese University-affiliated tertiary hospital (Mater Dei Hospital) under varying conditions, including varying light intensity, different patient positions and periods of time where clinical staff are performing regular care tasks and minor interventions such as bloodletting. Patients enrolled will be able to provide consent for the study after being given a detailed explanation of the study aims, data collected, data storage and processing and any other information they may wish to know.

The video data will be analysed via a convolutional neural network which has been previously trained to extract cardiovascular and respiratory parameters from videos taken from healthy volunteers in a non-clinical setting (a laboratory located in the University of Malta). The heart rate and respiratory rate extracted from patient videos are then compared to ground truth data obtained by current gold standard contact monitoring (data collected from Phillips Intellivue monitors used throughout the ICU) and assessed for accuracy. The practicality of setting up a camera-based system in the intensive care setting and potential means of overcoming limitations faced will also be tackled in this study from a qualitative aspect.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years and able to provide consent

Exclusion Criteria:

* age under 18 years and known cardiovascular or respiratory diseases

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients that fit into the inclusion criteria are included in the study regardless of underlying comorbidities or reasons for admission to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate as measured by a camera system | 1 day
Heart Rate, as measured by a camera system | 1 day

SECONDARY OUTCOMES:
To assess the accuracy of parameters obtained via the camera-based system as compared to the traditional contact monitoring system. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: Undecided